CLINICAL TRIAL: NCT02502084
Title: Safety and Effectiveness Evaluation of the Sinusway Device for Endoscopy of the Nasal Cavity and Paranasal Sinuses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3NT Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3NT-IL1
Record Dates: First submitted 2015-07-13; First posted 2015-07-20 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-01

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3NT flexible endoscope (Experimental): Evaluation of 3NT flexible endoscope in terms of access and evaluation of the nasal anatomy
  Interventions: Device: 3NT flexible endoscope

INTERVENTIONS:
Device: 3NT flexible endoscope — The nasal anatomy will be accessed and viewed with the device during functional endoscopic sinus surgery (FESS) procedure.
  Other Names: Sinusway

SUMMARY:
3NT flexible endoscope is a single-use disposable handheld endoscope that provides a means to visualize the nasal cavity and paranasal sinus space and deliver irrigation to treat the sinus ostia and spaces within the paranasal sinus cavities for diagnostic and therapeutic procedures.

DETAILED DESCRIPTION:
The rationale behind this feasibility study is to show that accessing and visualization of the nasal anatomy and paranasal sinuses (Maxillary, Frontal and Sphenoid sinuses) in patients suffering from symptoms attributable to sinusitis is feasible; This is an essential step in the development of a system that will later allow visualization, sampling, and treatment of the sinuses via the natural sinus ostium during the patient's first office visit in a minimally invasive manner while enabling treatment by lavage, and minimizing radiation exposure, antibiotic use, multiple office visits, and cost.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient indicated for primary FESS procedure by the ear, nose and throat (ENT) specialist
* Patient age: adult (>18 years old)
* Patients in general good health in the opinion of the investigator as determined by medical history physical examination
* A patient who is able to understand the requirements of the study, is willing to comply with its instructions and schedules, and agrees to sign the informed consent

Exclusion Criteria:

* A patient with nasal polyposis
* A patient indicated for tumor excision
* Known history of any significant medical disorder, which in the investigator's judgment contraindicates the patient's participation
* Patients with known current or previous bleeding disorder receiving anticoagulants (e.g., chronic Coumadin treatment)
* Pregnancy
* Patients with previous FESS surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety assessed by unanticipated device-related adverse events | During hospital stay, up to 1 day

SECONDARY OUTCOMES:
Performance assessed by anatomical landmarks reached and visualized will be recorded | During procedure, up to 3 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Ghent University, Ghent, Belgium
- Assuta Medical Center, Tel Aviv, Israel